CLINICAL TRIAL: NCT00120419
Title: Mycophenolate Mofetil in Antiretroviral Naïve Patients 2 (MAN2 Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanquin Research & Blood Bank Divisions (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAN2-study
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2006-01

CONDITIONS: HIV Infection
Keywords: HIV-1 infection; immunomodulatory therapy; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Mycophenolic Acid; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mycophenol mofetil (MMF, Cellcept®) 500 mg BID

SUMMARY:
The purpose of the study is to evaluate whether mycophenolate mofetil (MMF) can treat the chronic hyperactivation of the immune system and (partly) prevent the decrease of the CD4+ T-cell count in chronically HIV-1 infected patients who are not treated with antiretroviral therapy (ART). The researchers also want to know what the effect is of treatment with MMF on plasma HIV-1 RNA; progression of disease (occurrence of AIDS defining events or reaching the indication to start ART); and the safety of treatment with MMF in this patient group.

DETAILED DESCRIPTION:
*Background: During chronic HIV-1 infection the immune system is chronically hyperactivated. This hyperactivation is considered as the main cause of CD4+ T-cell loss. Furthermore, HIV replicates most efficiently in activated CD4+ T-cells. In this study we try to inhibit the activation of the immune system with mycophenolate mofetil (MMF). Previous studies in which HIV-1 infected patients have been treated with MMF in addition to antiretroviral treatment (ART) have not shown any additional effect, compared to ART alone. In this study MMF will be used without antiretroviral medication.

*Objectives: Primary objective of the study is the evaluation of the effect of MMF on the chronic hyperactivation of the immune system and the decrease of the CD4+ T-cell count in chronically HIV-1 infected patients who are not treated with antiretroviral therapy (ART). Secondary objectives include the evaluation of the effect of MMF on plasma HIV-1 RNA; progression of disease/ reaching of indication to start ART; and the safety of treatment with MMF in this patient group.

*Study Design: This is a multi center, randomized, open-label study, in which patients will be randomized to treatment with mycophenolate mofetil (MMF) 500 mg BID during 48 weeks versus no treatment. In a subgroup of 20 patients ("immunology group", the first 20 patients in the AMC hospital, Amsterdam, the Netherlands) a number of additional immunological measurements will be performed.

The study duration is 60 weeks (48 weeks of treatments with 1 additional visit 12 weeks after cessation of treatment).

*Study Population: Potential participants are adult chronically HIV-1 infected patients, who have never been treated with ART and who according to the present criteria do not need to be treated. CD4+ T lymphocyte count has to be > 250 and <= 450 * 106/L, plasma HIV-1 RNA (viral load) < 10.000 copies/ mL.

*Intervention: Patients will be randomized (1:1) to mycofenolate mofetil (MMF) 500 mg BID versus no treatment.

*Endpoints: Primary endpoints are change over time (baseline - week 48) in CD4+ T cell count and peripheral blood lymphocyte (PBMC) activation markers.

Secondary endpoints are changes over time (baseline - week 48) in plasma HIV-1 RNA, time to reach indication to start ART (separated in three groups: 1. two consecutive measurements of CD4+ T cell count below 250 * 106 cells/ L with at least 4 weeks interval; 2. the occurrence of a CDC class B or C event; 3. any other reason); safety data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age;
* Patient has a proven HIV-1 infection (with antibodies against HIV-1 and a detectable plasma HIV-1 RNA measured for the first time at least 6 months prior to inclusion);
* Patient is HIV-1 treatment naïve;
* CD4+ T lymphocyte count > 250 and <= 450 * 106/L;
* No signs or history of AIDS defining events;
* No use of other medications that might possibly influence the effects of MMF;
* Male; or female sex and willingness to practice effective contraception during the study.

Exclusion Criteria:

* Plasma HIV-1 RNA < 10.000 copies/ mL;
* Autoimmune disease;
* Active hepatitis B or C virus infection;
* Other chronic diseases;
* Recent infectious disease other than HIV-1;
* Treatment with immunomodulatory or anti-inflammatory medication in the past 6 months;
* For female patients: pregnancy and lactation;
* Any other condition, illness or use of medication which according to the investigator is not compatible with the use of the study medication or which could interfere with the evaluations required by the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-04

PRIMARY OUTCOMES:
Change over time (baseline - week 48) in CD4+ cell counts in peripheral blood and peripheral blood lymphocyte activation markers.

SECONDARY OUTCOMES:
* Change over time (baseline - week 48) in plasma HIV-1 RNA, time to reach an indication to start antiretroviral treatment and safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Prins, MD PhD, Principal Investigator — Department of Internal Medicine, Division of Infectious Diseases, Tropical Medicine and AIDS, Academic Medical Center, University of Amsterdam, the Netherlands; Kees Brinkman, MD PhD, Principal Investigator — department of internal medicine, OLVG hospital, Amsterdam, the Netherlands; Robin Soetekouw, MD, Principal Investigator — department of internal medicine, Kennemer Gasthuis, Haarlem, the Netherlands; Robert Kauffmann, MD PhD, Principal Investigator — Department of Internal Medicine, HAGA hospital, location Leyenburg Hospital, The Hague, The Netherlands
Locations (5):
- Netherlands (5):
  - OLVG, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - Kennemer Gasthuis, location EG, Haarlem, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - HAGA hospital, location Leyenburg Hospital, The Hague, South Holland

REFERENCES:
- [Background] Chapuis AG, Paolo Rizzardi G, D'Agostino C, Attinger A, Knabenhans C, Fleury S, Acha-Orbea H, Pantaleo G. Effects of mycophenolic acid on human immunodeficiency virus infection in vitro and in vivo. Nat Med. 2000 Jul;6(7):762-8. doi: 10.1038/77489. PMID 10888924
- [Background] Sankatsing SU, Jurriaans S, van Swieten P, van Leth F, Cornelissen M, Miedema F, Lange JM, Schuitemaker H, Prins JM. Highly active antiretroviral therapy with or without mycophenolate mofetil in treatment-naive HIV-1 patients. AIDS. 2004 Sep 24;18(14):1925-31. doi: 10.1097/00002030-200409240-00008. PMID 15353978
- [Background] Garcia F, Plana M, Arnedo M, Brunet M, Castro P, Gil C, Vidal E, Millan O, Lopez A, Martorell J, Fumero E, Miro JM, Alcami J, Pumarola T, Gallart T, Gatell JM. Effect of mycophenolate mofetil on immune response and plasma and lymphatic tissue viral load during and after interruption of highly active antiretroviral therapy for patients with chronic HIV infection: a randomized pilot study. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):823-30. doi: 10.1097/00126334-200407010-00009. PMID 15213566